CLINICAL TRIAL: NCT06600217
Title: Développement De La Stimulation Non-invasive En Boucle Fermée
Brief Title: Closed-loop Non-invasive Brain Stiumlation
Acronym: CLOSEDLOOP
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Collaborators: Laboratoire de Psychologie et NeuroCognition (LPNC), UniversitÃ© Grenoble Alpes (Unknown); GIPSA-lab, Grenoble, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 38RC24.0193; 2024-A01226-41 (Other: ID-RCB)
Record Dates: First submitted 2024-09-12; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Non-invasive Brain Stimulation; Methodologic Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy subjects

SUMMARY:
Transcranial magnetic stimulation (TMS) is a widely used tool for exploring brain function in humans (Siebner et al. et al., 2022), which has led to new therapeutics for various psychiatric and neurological disorders (Lefaucheur et al., 2020). However, the open-loop use of this technique has raised questions about its operating principle, due to the high degree of heterogeneity of results and the small to medium observed effect sizes (Zrenner and Ziemann, 2023). To increase the response rate, it has been suggested to individualize stimulation, by adapting the TMS parameters (i.e. delivered dose, target dose, targeting, timing, etc.) to instantaneous estimates of brain brain state. Such an approach, known as closed-loop closed-loop stimulation, is currently one of the main challenges challenges in this field (closed-loop brain state-dependent stimulation). To this end, we are focusing on the combination of robotic TMS and electroencephalography (EEG) (Hernandez-Pavon et al. al., 2023). The closed-loop stimulations using this combination developed to date have two limitations: (i) they are not adaptive and focus focus mainly on calculating the phase of brain oscillations to trigger stimulation and (ii) are limited to central cortical (sensorimotor) areas, where the EEG signal-to-noise ratio is optimal.

This project aims to develop closed-loop TMS-EEG protocols that overcome these two limitations: (i) by incorporating adaptive decision modeling (AutoHS model, Harquel et al. 2017) to optimize several parameters in parallel (coil location, orientation, intensity) while using a wider range of EEG markers (evoked potentials, oscillatory activity strength, connectivity, etc.), and (ii) by integrating real-time EEG pre-processing to access any cortical target (including frontal, temporal and occipital lobes).

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Having undergone a medical examination prior to participation in research
* Affiliation with or beneficiary of a social security scheme

Exclusion Criteria:

* Contraindications (CI) to MRI, EEG, TMS practice
* Existence of a severe general medical condition: cardiac, respiratory, hematological, renal, hepatic, cancerous,
* Regular use of anxiolytics, sedatives, antidepressants, neuroleptics,
* Characterized psychiatric pathology,
* Suspicion of alcohol ingestion prior to the examination,
* Participation in other interventional research protocols in progress with exclusion period or in the preceding week.
* Persons covered by articles L1121-5 to L1121-8 of the CSP (French Public Health Code) (corresponds to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, persons under psychiatric care under articles L.

3212-1 and L. 3213-1 who are not covered by the provisions of article L. 1121-8, persons admitted to a health or social establishment for purposes other than research, minors, persons under legal protection or unable to express their consent).

- Personnel with a hierarchical link to the principal investigator

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy volunteers from Grenoble and the surrounding area
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Quality of EEG markers extracted in real-time | During the two TMS-EEG experimental sessions, at day 0 and up to day 30
  Quality of EEG markers extracted in real-time (evoked potentials, power and phase of brain oscillations and functional connectivity)
Quality of EEG marker modulation | During the two TMS-EEG experimental sessions, at day 0 and up to day 30
  Quality of EEG marker modulation induced by TMS parameters selected by the AutoHS decision model

SECONDARY OUTCOMES:
Intra-individual (inter-session) reproducibility of primary endpoint quality markers | Contrast between the 2 TMS-EEG experimental sessions, at day 0 up to day 30
  Intra-individual (inter-session) reproducibility of primary endpoint quality markers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harquel S, Diard J, Raffin E, Passera B, Dall'Igna G, Marendaz C, David O, Chauvin A. Automatized set-up procedure for transcranial magnetic stimulation protocols. Neuroimage. 2017 Jun;153:307-318. doi: 10.1016/j.neuroimage.2017.04.001. Epub 2017 Apr 5. PMID 28389385